CLINICAL TRIAL: NCT03696394
Title: A Pilot Study to Evaluate the Efficacy of BioCartilage® Micronized Cartilage Matrix in Microfracture Treatment of Osteochondral Defects of the Talus
Brief Title: A Study to Evaluate the Efficacy of BioCartilage® Micronized Cartilage Matrix in Microfracture Treatment of Osteochondral Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Paul's Hospital, Canada (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Principal Investigator, Andrea Veljkovic, Orthopaedic Surgeon, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ART - BioCartilage; H18-00603 (Other: UBC Providence Health Care Research Ethics Board)
Record Dates: First submitted 2018-10-01; First posted 2018-10-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Osteochondral Defect

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups. Group I consists of 5 patients receiving Microfracture as per standard of care (Control Group). Group II consists of 10 patients receiving Microfracture with BioCartilage® (Investigational Group).
Who Masked: Participant
Masking Description: This study will be single-blinded. Group I and II subjects will be blinded as to whether they have received BioCartilage® in addition to Microfracture or Microfracture alone, as per standard of care. Investigators will be aware of the assigned treatment on the patients. Subjects will be aware of their assigned treatment after their surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (No Intervention): Group I consists of 5 patients receiving a microfracture as per standard of care.
- Group II (Active Comparator): Group II consists of 10 patients receiving a microfracture with BioCartilage®.
  Interventions: Device: BioCartilage® Micronized Cartilage Matrix

INTERVENTIONS:
Device: BioCartilage® Micronized Cartilage Matrix — BioCartilage® is a scaffold with Collagen Type II and cartilage matrix elements
  Other Names: BioCartilage®
  Arms: Group II

SUMMARY:
The study was designed by the principal investigator, Dr. Andrea Veljkovic, and the St. Paul's Hospital Foot and Ankle Research Group, who will conduct the study. The study is being funded by Arthrex, Inc., the manufacturer of the Health Canada approved BioCartilage® Micronized Cartilage Matrix.

The purpose of this study is to assess whether adding BioCartilage® to microfracture treatment of osteochondral defects of the talus improves osteochondral healing as well as improving pain and function.

Efficacy will be assessed primarily by outcomes scores as measure by the Ankle Osteoarthritis Scale (AOS) at the baseline and at multiple post-op followup visits. Additional outcomes scores will also be administered to compare general health and foot function between the two groups at baseline and at multiple post-op followup visits. X-rays and MRI will be used to assess the osteochondral healing rate.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has signed the REB approved informed consent form (ICF) specific to this study prior to enrollment.
2. The subject has an isolated OCD with minimum dimensions of 0.07 cm2 (0.3 cm in diameter) and maximum dimensions of 2.25 cm2 as confirmed by a pre-op MRI.
3. The subject is independent, ambulatory, and can comply with all post-operative evaluations and visits.
4. The subject is at least nineteen (19) years of age and considered to be skeletally mature.
5. The subject has a combined bone and cartilage defect as determined by an MRI.
6. The patient has a stable ankle joint on history and has similar ligament stability with the opposite ankle.
7. The subject has less than 15 degrees of hindfoot valgus and 5 degrees of hindfoot varus.
8. The subject has a chronic defect not secondary to acute trauma within the last 6 months.
9. The patient (if having suffered a fracture) has no residual deformity of the tibia, fibula or syndesmosis.
10. The subject has a BMI of ≤ 40 kg/m².
11. The subject has exhausted non-operative treatment.
12. The subject has symptoms for less than a year.
13. Lesions on the subject must be contained.

Exclusion Criteria:

1. The subject has over 15 degrees of hindfoot valgus or 5 degrees of hindfoot varus.
2. The subject has an isolated OCD with dimensions greater than 2.0 cm2 on an MRI assessment.
3. The subject has an allergy to yeast-derived products.
4. The subject has implanted metallic devices (cardiac pacemakers, insulin pumps, and nerve stimulators), medically implanted clips, or other electronically, magnetically or mechanically activated implants that would contraindicate an MRI scan of the foot.
5. The subject has claustrophobia that would inhibit their ability to undergo an MRI scan of the foot.
6. The subject has tested positive or has been treated for a malignancy in the past, is suspected of having a malignancy, or is currently undergoing radiation or chemotherapy treatment for a malignancy anywhere in the body, whether adjacent to or distant from the proposed BioCartilage® site.
7. The subject is physically or mentally compromised (e.g., currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, etc.), to the extent that the investigator judges the subject to be unable or unlikely to remain compliant to follow-up.
8. The subject is a prisoner, or is known or suspected to be transient.
9. The subject has documented evidence of a history (e.g. liver testing) of drug/alcohol abuse within the 12 months prior to screening for study entry.
10. The subject is pregnant or able to become pregnant but not practicing a medically-accepted form of birth control, and/or intending to become pregnant during this study period.
11. The subject currently has an acute infection in the area surrounding the surgical site.
12. The subject has a history of anaphylaxis or of multiple non-environmental allergies that may precipitate an anaphylactic reaction.
13. The subject's condition is bilateral and surgery is scheduled or to be scheduled over the course of this trial for both feet.
14. The subject requires a concomitant osteotomy of the tibia, fibula, or calcaneus for hindfoot deformity.
15. The subject requires a concomitant hindfoot fusion or has had a hindfoot fusion for hindfoot arthritis or deformity.
16. The subject is undergoing any concomitant surgery that may invalidate the outcome scores such as forefoot surgery or fusions, tendon transfers or ligament reconstructions. Heel cord lengthening is permitted.
17. The subject has an OCD of the tibia in isolation or in combination with the talar lesion
18. The subject is addicted to nicotine and on nicotine containing medication such as gum or a patch; or using nicotine containing substances such as cigarettes, cigars, pipe smoking or chewing tobacco.
19. The subject abuses cocaine or cocaine derivative drugs.
20. The subject has a known hypersensitivity to aprotinin.
21. The subject has diabetes with an HBA1c> 7.5.
22. The subject is unable to give informed consent.
23. The subject is unable to comply with follow-up.
24. The subject is unable to communicate with the research team.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Changes as Assessed by Ankle Osteoarthritis Scale (AOS) | Outcome will be administered 6 times per patient: within 21 days of surgery, 6 weeks post-op, 12 weeks post-op, 6 months post-op, 1 year post-op and 2 years post-op.
  This questionnaire assesses pain and difficulty in both the left and right ankle. The range for the Pain subscale is from 0 to 100 and the range for the Difficulty subscale is 0 to 100. The range for the Total score (average of Pain and Difficulty) is 0 to 100. Lower values for Pain, Difficulty, and Total is considered better.
  The scores will be compared to each other to analyze the change in pain and difficulty from the baseline (within 21 days of surgery) to the end (2 years post-op).

SECONDARY OUTCOMES:
Musculoskeletal Outcomes Data Evaluation and Management System (MODEMS) including Short Form 36 Health Survey (SF-36) | Outcome will be administered 6 times per patient: within 21 days of surgery, 6 weeks post-op, 12 weeks post-op, 6 months post-op, 1 year post-op and 2 years post-op.
  This questionnaire assesses multiple aspects patient health such as comorbidities, expectations/satisfaction, physical component score and mental component score. These measures and scores are values on a unitless scale.
Foot and Ankle Ability Measure (FAAM) | Outcome will be administered 6 times per patient: within 21 days of surgery, 6 weeks post-op, 12 weeks post-op, 6 months post-op, 1 year post-op and 2 years post-op.
  This questionnaire assesses activities of daily living and sports subscales. Both subscales range from "Unable to Do", which indicates a minimum score of 0, to "No Difficulty", which indicates a maximum score of 4. A better outcome would be a higher score for both subscales.
  There is one last questions which asks the patient about their current level of function during their usual activities of daily living (daily living subscale) and sports (sports subscale). For both subscales, the range is from a minimum of 0% to a maximum of 100%. A better outcome score would be a higher score for both subscales.
  Both of these subscales are not combined to compute a total score.
Visual Analog Scale | Outcome will be administered 6 times per patient: within 21 days of surgery, 6 weeks post-op, 12 weeks post-op, 6 months post-op, 1 year post-op and 2 years post-op.
  This questionnaire assesses the current level of pain in the foot/ankle that was treated. This scale ranges from "No Pain", which indicates a minimum score of 0, to "Worst Pain", which indicates a maximum score of 10. A better outcome would be a lower score.
X-ray radiographic assessments performed pre-operatively and post-operatively | There are 6 assessment time points: within 21 days of surgery, 6 weeks post-op, 12 weeks post-op, 6 months post-op, 1 year post-op and 2 years post-op.
  X-rays will be completed to assess osteochondral healing.
CT radiographic assessments performed pre-operatively and post-operatively | There are 2 assessment time points: within 21 days of surgery and 2 years post-op.
  CTs will be completed to assess osteochondral healing.
MRI radiographic assessments performed pre-operatively and post-operatively | There are 2 assessment time points: within 21 days of surgery and 2 years post-op.
  MRIs will be completed to assess osteochondral healing.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No